CLINICAL TRIAL: NCT05336578
Title: Comparative Investigation of Anti-inflammatory Effect of Platelet-Rıch Fıbrın After Mandibular Wisdom Tooth Surgery
Brief Title: Anti-inflammatory Effect of Platelet-Rıch Fıbrın
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nilay Er (Other)
Responsible Party: Sponsor-Investigator, Nilay Er, Assistant Professor, Trakya University
Organization: Trakya University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: PRF2022
Record Dates: First submitted 2022-04-06; First posted 2022-04-20 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Surgical Complication; Pain, Postoperative; Edema Face
Keywords: platelet-rich-fibrin; edema; Serum markers; trismus
MeSH Terms: conditions — Pain, Postoperative; Edema; Trismus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1- PRF (Experimental): After wisdom tooth extraction PRF located to the extraction socket
  Interventions: Other: Platelet rich fibrin application
- PRF free (No Intervention): Only surgical procedure of the wisdom tooth extraction is performed

INTERVENTIONS:
Other: Platelet rich fibrin application — PRFs were prepared by obtaining10 ml blood samples from each patinet and inserting them in a centrifuge device (Intra-Lock International Inc., Boca Raton, USA), under 2700 rpm for 12 min using high speed. The platelet-rich fibrin layer remaining between the acellular plasma and red blood cells in the tube was separated with the help of scissors or a scalpel. After the tooth extraction in the experimental group PRF located to the extraction socket.
  Arms: 1- PRF

SUMMARY:
This study evaluated the anti-inflammatory effect of platelet-rich fibrin (PRF) applied to the extraction socket after impacted mandibular third molar surgery with subjective and objective parameters. A total of 48 patients who had fully impacted wisdom teeth in bilateral and similar positions were included in the study. The control group was formed with the standard extraction of the lower third molars, and the PRF group was formed with local PRF application in addition to standard impacted tooth surgery (n=96). The anti-inflammatory activity of PRF on postoperative 2nd and 7th days was evaluated subjectively by clinical parameters and objectively by biochemical parameters.

Subjective parameters were pain assesment, swelling measurements on the face and limitation of mouth opening. Objective data is the analysis of serum values and anti-inflammatory markers in the blood.

DETAILED DESCRIPTION:
Operations All surgical procedures were performed by the same surgeon, with the same flap design and the same surgical technique. 2 ml of a local anesthetic solution containing 40 mg/ml articaine HCl and 0.006 mg/ml epinephrine HCl was used for N. alveolaris inferior and N. buccalis blockage. The mucoperiosteal flap was removed by making a horizontal incision starting from the retromolar region, through horizontally in the buccal, circular around the neck of the mandibular second molar, and continuing vertically at the mesial half of the mandibular second molar tooth. Alveolotomy and/or division of teeth and/or roots were performed with sterile tungsten carbide burs with an electric controlled motor rotating at 20,000 rpm under 0.9% saline irrigation during operation. Roots were removed from the alveoli with the help of a bein elevator placed on the buccal and/or mesial parts of the teeth. After tooth extraction, the bone, soft tissue residues, and debris in the area were removed, and the socket was irrigated with 0.9% saline. In the control group, primary suturing was performed after bleeding control without any application to the extraction socket, while in the PRF group, PRF was applied to the socket just before suturing (Fig 2). All patients were prescribed antibiotics (amoxicillin-clavulanic acid, 1gr, 2x1) (Augmentin-BID, GlaxoSmithKline, London, England), analgesic (Acetaminophen, 500 mg, 3x1) (Parol, Atabay, Istanbul, Turkey) and mouthwash (120 mg %0.12 chlorhexidine gluconate and 150 mg %0.15 benzydamine hydrochloride, 200 ml, 3x1) (Kloroben, Drogsan, Ankara, Turkey) after the surgical procedure.

PRF Preparation Blood sampling was performed through the peripheral antecubital vein by selecting a suitable branule for the patient's vascular structure with a closed vacuum system. PRFs were prepared according to the method of Choukron et al.(2001). 10 ml blood samples were inserted in a centrifuge device (Intra-Lock International Inc., Boca Raton, USA), under 2700 rpm for 12 min using high speed. The platelet-rich fibrin layer remaining between the acellular plasma and red blood cells in the tube was separated with the help of scissors or a scalpel.

Obtaining edema, pain, and serum marker data A visual analog scale (VAS) of 100 mm was given to the patients to determine the severity of pain on the operation day and on the 2nd and 7th postoperative days, with 0 indicating no pain and 100 indicating the worst pain they had ever experienced. In order to evaluate the severity of edema, the tragus - buccal comissura and lateral canthus - gonion distances of the patients were measured using a flexible ruler before the operation and on the 2nd and 7th days postoperatively, and the results were recorded. To evaluate the trismus level, the interincisal distance of the patients was measured with a flexible ruler before the operation and on the 2nd and 7th days postoperatively in both groups. The progression of swelling and trismus was measured in millimeters and evaluated by comparing with the value obtained at baseline14.

For objective data, ESR values were measured using the Vision ESR analyzer (YHLO Biotech Co., Shenzhen, China), and CRP values were measured using the BN II nephelometric analyzer (Siemens Healthcare Diagnostics, Marburg, Germany). IL-6 levels (pg/ml) were determined using the Human IL-6 Elisa Kit (Elabscience Biotechnology Co., Wuhan, China) and TNF-a levels (pg/ml) were determined using the Human TNF-α Elisa Kit (Elabscience Biotechnology Co., was measured using Wuhan, China).

Statistical Evaluation Data were analyzed with the IBM SPSS® V23 (IBM Company, Chicago, IL, United States) package program. Mann-Whitney U test was used to compare non-normally distributed data according to paired groups, and an independent two-sample t-test was used to compare normally distributed data. The significance level was taken as p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* not have any systemic disease that will prevent tissue healing
* no history of regular drug use
* no drug allergies
* not smoking
* not being pregnant
* having bilateral mandibular third molar tooth in class II, position B and C position according to Pell & Gregory classification with the same root form, position and level of impaction
* no signs of abscess, pericoronitis or inflammation before extraction

Exclusion Criteria:

* pregnancy
* having a chronic disease
* having a local infection in the impacted tooth area
* smoking

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2020-02-10 (Actual); Study Completion 2021-08-22 (Actual)

PRIMARY OUTCOMES:
Edema measurement | 2nd day posoperatively
  In order to evaluate the severity of edema, the tragus - mouth corner and lateral canthus - gonion distances of the patients were measured using a flexible ruler before the operation and on the 2nd and 7th days postoperatively, and the results were recorded.
Edema measurement | 7th day posoperatively
  In order to evaluate the severity of edema, the tragus - mouth corner and lateral canthus - gonion distances of the patients were measured using a flexible ruler before the operation and on the 2nd and 7th days postoperatively, and the results were recorded.
Trismus measurement | 2nd day postoperatively
  To evaluate the trismus level, the interincisal distance of the patients was measured with a flexible ruler before the operation and on the 2nd and 7th days postoperatively in both groups.
Trismus measurement | 7th day postoperatively
  To evaluate the trismus level, the interincisal distance of the patients was measured with a flexible ruler before the operation and on the 2nd and 7th days postoperatively in both groups.
Pain assesment | 2nd day postoperatively
  A visual analog scale (VAS) (Validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain") was given to the patients to determine the severity of pain on the operation day and on the 2nd and 7th postoperative days.
Pain assesment | 7th day postoperatively
  A visual analog scale (VAS) (Validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain") was given to the patients to determine the severity of pain on the operation day and on the 2nd and 7th postoperative days.
Erythrocyte sedimentation rate (ESR) | 2nd day postoperatively
  A serum marker for analysing acute phase response, as it is necessary for initiating the inflammatory response
Erythrocyte sedimentation rate (ESR) | 7th day postoperatively
  A serum marker for analysing acute phase response, as it is necessary for initiating the inflammatory response
C-reactive protein (CRP) | 2nd day postoperatively
  A serum marker for analysing acute phase response, as it is necessary for initiating the inflammatory response
C-reactive protein (CRP) | 7th day postoperatively
  A serum marker for analysing acute phase response, as it is necessary for initiating the inflammatory response
interleukin 6 (IL-6) | 2nd day postoperatively
  A serum marker for analysing acute phase response, as it is necessary for initiating the inflammatory response
interleukin 6 (IL-6) | 7th day postoperatively
  A serum marker for analysing acute phase response, as it is necessary for initiating the inflammatory response
tumor necrosis factor-alpha (TNF-α ) | 2nd day postoperatively
  A serum marker for analysing acute phase response, as it is necessary for initiating the inflammatory response
tumor necrosis factor-alpha (TNF-α ) | 7th day postoperatively
  A serum marker for analysing acute phase response, as it is necessary for initiating the inflammatory response

CONTACTS AND LOCATIONS:
Overall Officials: Nilay Er, Principal Investigator — Trakya University
Locations (1):
- Trakya University, Edirne, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Del Corso M, Vervelle A, Simonpieri A, Jimbo R, Inchingolo F, Sammartino G, Dohan Ehrenfest DM. Current knowledge and perspectives for the use of platelet-rich plasma (PRP) and platelet-rich fibrin (PRF) in oral and maxillofacial surgery part 1: Periodontal and dentoalveolar surgery. Curr Pharm Biotechnol. 2012 Jun;13(7):1207-30. doi: 10.2174/138920112800624391. PMID 21740371
- [Result] Dar MM, Shah AA, Najar AL, Younis M, Kapoor M, Dar JI. Healing Potential of Platelet Rich Fibrin in Impacted Mandibular Third Molar Extraction Sockets. Ann Maxillofac Surg. 2018 Jul-Dec;8(2):206-213. doi: 10.4103/ams.ams_181_18. PMID 30693233
- [Result] Ozgul O, Senses F, Er N, Tekin U, Tuz HH, Alkan A, Kocyigit ID, Atil F. Efficacy of platelet rich fibrin in the reduction of the pain and swelling after impacted third molar surgery: randomized multicenter split-mouth clinical trial. Head Face Med. 2015 Nov 26;11:37. doi: 10.1186/s13005-015-0094-5. PMID 26607842
- [Result] Litao MK, Kamat D. Erythrocyte sedimentation rate and C-reactive protein: how best to use them in clinical practice. Pediatr Ann. 2014 Oct;43(10):417-20. doi: 10.3928/00904481-20140924-10. PMID 25290132
- [Result] Sahibzada HA, Khurshid Z, Khan RS, Naseem M, Siddique KM, Mali M, Zafar MS. Salivary IL-8, IL-6 and TNF-alpha as Potential Diagnostic Biomarkers for Oral Cancer. Diagnostics (Basel). 2017 Apr 9;7(2):21. doi: 10.3390/diagnostics7020021. PMID 28397778